CLINICAL TRIAL: NCT06901765
Title: Effectiveness of Kinesio Taping in Patients with Congenital Muscular Torticollis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sisli Hamidiye Etfal Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Aylin Ayyıldız, MD, Başakşehir Çam & Sakura City Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: KAEK-11/12.02.2025.52
Record Dates: First submitted 2025-03-23; First posted 2025-03-30 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Torticollis Congenital
MeSH Terms: conditions — Congenital torticollis | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Research Group (Active Comparator): In addition to the regular exercise program, patients diagnosed with Congenital Muscular Torticollis will be given kinesio taping for torticollis. Kinesio taping will be applied for 4 weeks, with 5 days on and 2 days off.
  Interventions: Procedure: Kinesiotaping; Behavioral: Exercise
- Control Group (Sham Comparator): Patients diagnosed with Congenital Muscular Torticollis will continue their regular exercise program. No intervention will be applied.
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Procedure: Kinesiotaping — Kinesio Taping Method is a therapeutic tool utilised by rehabilitation specialists in all programs (paediatric, geriatric, orthopaedic, neurological, oncology and others) and levels of care (acute care, inpatient rehabilitation, outpatient, home care and Day Rehab). The idea of using elastic tape to mimic the therapist's hands was first presented by Dr Kenzo Kase in the 1970s. Since then, it became the modality used in pain management[5], soft tissue injury, tissues and joints malalignment, oedema, and more. Kinesio Taping Method utilises four types of Kinesio Tex Tapes, each with specific properties designed for use on fragile, sensitive skin or applied with higher tensions. Kinesio Taping Method has also effectively treated animals and two special tapes are used: Kinesio Equine and Kinesio Canine. Kinesio Tex Tape contains either 100% cotton and elastic fibres or a blend of polyester and cotton with elastic fibres. The latter is preferable for Kinesio Taping application on sensitive
  Arms: Research Group
Behavioral: Exercise — Range of Motion Exercise, Stretching Exercises

SUMMARY:
The aim is to investigate the effectiveness of kinesiotaping application in addition to Congenital Muscular Torticollis exercise on neck joint range of motion, tilt degree and muscle function test. Research Group: In addition to the regular exercise program, patients diagnosed with Congenital Muscular Torticollis will be given kinesio taping for torticollis. Kinesio taping will be applied for 4 weeks, 5 days on and 2 days off. Control Group: Patients diagnosed with Congenital Muscular Torticollis will continue their regular exercise program. No intervention will be applied. Patients will be evaluated with neck joint range of motion, tilt degree and muscle function test before and 3 months after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Being followed up with a diagnosis of Congenital Muscular Torticollis
* The family's willingness to participate in the study

Exclusion Criteria:

* Presence of cardiopulmonary disease and musculoskeletal deformity that will prevent exercise
* Having an open wound in the area where kinesio taping will be applied or being allergic to tape application

Ages: 0 Years to 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 54 (Estimated)
Dates: Start 2025-03-28 (Estimated); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Range of Motion Measurement | 3 months
tilt degree | 3 months

SECONDARY OUTCOMES:
Muscle Function Scale | 3 months